CLINICAL TRIAL: NCT07269067
Title: Multicenter Retrospective Cohort Assessing Concordance Between Manual Gating and Unsupervised FlowSOM Gating for Minimal Residual Disease Detection by Multiparameter Flow Cytometry in Adult and Paediatric Acute Myeloid Leukaemia
Brief Title: Automated vs Manual Flow-cytometry Gating for Measurable Residual Disease in Acute Myeloid Leukaemia (DUALFLOW)
Acronym: DUALFLOW
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2025/033
Record Dates: First submitted 2025-11-21; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Acute Myeloid Leukemia; Minimal Residual Disease; Flow Cytometry; FlowSOM; Gating Algorithm; Machine Learning
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adult AML cohort: Adults ≥ 18 years with ELN-defined AML enrolled in DATAML Bordeaux, possessing flow-cytometry MRD data after induction and consolidation 1
  Interventions: Diagnostic Test: Conventional gating; Diagnostic Test: Automated gating
- Paediatric AML cohort: Children and adolescents 0-18 years managed in the paediatric haemato-oncology unit, with analogous MRD flow-cytometry data
  Interventions: Diagnostic Test: Conventional gating; Diagnostic Test: Automated gating

INTERVENTIONS:
Diagnostic Test: Conventional gating — Manual expert gating of multiparameter flow-cytometry data for MRD
Diagnostic Test: Automated gating — Unsupervised FlowSOM gating of multiparameter flow-cytometry data for MRD

SUMMARY:
This retrospective multicentre cohort evaluates the agreement of measurable residual disease (MRD) detection in acute myeloid leukaemia (AML) using two flow-cytometry gating approaches. Manual expert gating is compared with an unsupervised FlowSOM clustering algorithm across post-induction and post-consolidation samples from 50 adults and 10 paediatric patients treated at Bordeaux University Hospital. The primary hypothesis states that unsupervised gating detects MRD ≥ 0.1 % with sensitivity and specificity comparable to manual gating.

DETAILED DESCRIPTION:
Acute myeloid leukaemia remains associated with high relapse rates despite complete remission after induction chemotherapy. Sensitive identification of residual leukaemic blasts (MRD) guides risk-adapted therapy. Flow cytometry is applicable to nearly all patients but relies on operator-dependent manual gating, which may lack reproducibility when rare or immunophenotypically atypical blasts are present. A data-driven alternative based on FlowSOM clustering was developed at Bordeaux to overcome these limitations. DualFlow retrospectively analyses paired flow-cytometry standard (FCS) files from 60 AML patients (≈ 100 MRD determinations) drawn from the DATAML Bordeaux adult database and the paediatric haemato-oncology service. Files are distributed to three partner centers for blinded re-analysis. Each sample undergoes: (1) conventional manual gating in two expert centers; (2) unsupervised FlowSOM gating in one center; (3) molecular MRD assessment when available. Primary analysis calculates sensitivity, specificity, predictive values and Cohen/Fleiss kappa for MRD ≥ 0.1 %. Secondary analyses include concordance with molecular MRD, Bland-Altman and correlation for MRD 0.01-0.1 %, impact on relapse-free and overall survival using Kaplan-Meier and Cox models, and operator reproducibility for manual gating. Covariate effects (age, cytogenetics, molecular risk, treatment) are explored through stratified and multivariable methods. No additional interventions or specimens are collected; only de-identified FCS files and routine clinical data are used.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of acute myeloid leukaemia per ELN 2022
* Age ≥ 18 years (adult cohort) or 0-20 years (paediatric cohort)
* Inclusion in DATAML Bordeaux database or paediatric haemato-oncology records
* Available flow-cytometry MRD data post-induction and post-consolidation 1
* Non-opposition or consent for secondary use of data

Exclusion Criteria:

* AML subtypes M3, M6 or M7
* Acute leukaemia of ambiguous lineage
* Missing or unusable flow-cytometry files for required time points

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive adult and paediatric patients diagnosed with ELN-defined AML at Bordeaux University Hospital between 2010 and 2024, for whom routine multiparameter flow-cytometry MRD assessments post-induction and post-consolidation 1 are available
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Concordance of MRD ≥ 0.1 % between manual gating and unsupervised FlowSOM gating | up to 8 weeks after initiation first cycle of intensive therapy and after initiation of second cycle of intensive therapy
  Sensitivity, specificity, positive and negative predictive values, Cohen and Fleiss kappa statistics comparing the 3 methods on paired samples

SECONDARY OUTCOMES:
Concordance of flow-cytometry MRD (both methods) with molecular MRD | up to 8 weeks after initiation first cycle of intensive therapy and after initiation of second cycle of intensive therapy
  Sensitivity, specificity, positive and negative predictive values, Cohen and Fleiss kappa statistics comparing the 3 methods on paired samples
Agreement of MRD 0.01-0.1 % between manual and unsupervised gating | up to 8 weeks after initiation first cycle of intensive therapy and after initiation of second cycle of intensive therapy
  Bland-Altman limits of agreement and Pearson or Spearman correlation coefficients calculated from log-transformed MRD percentages to assess agreement between both gating methods in the low MRD range
Concordance of flow-cytometry MRD (both methods) with molecular MRD | From diagnosis up to 60 months
  Kaplan-Meier survival analyses and multivariable Cox regression models used to compare relapse-free survival (RFS) and overall survival (OS) according to MRD detection method
Inter-operator reproducibility of manual gating | up to 8 weeks after initiation first cycle of intensive therapy and after initiation of second cycle of intensive therapy
  Intra-class correlation coefficients and Fleiss kappa statistics calculated across three independent operators performing manual gating on the same flow-cytometry MRD files

IPD SHARING:
Plan to Share IPD: No